CLINICAL TRIAL: NCT03546439
Title: VAscular Closure for Cardiac Ablation Registry (VACCAR)
Acronym: VACCAR
Status: Completed | Type: Observational
Sponsor: Saint Luke's Health System (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: VACCAR
Record Dates: First submitted 2018-05-21; First posted 2018-06-06 (Actual); Results first posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2021-12

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; vascular closure
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this registry is to find out if there is a difference in patient satisfaction and rate of vascular and bleeding complications with use of Perclose Proglide system or F08S for venous closure post atrial fibrillation and atrial flutter procedures in comparison to manual compression.

DETAILED DESCRIPTION:
Vascular Closure Devices (VCD) have been used to achieve hemostasis of arterial access sites following cardiac catheterization procedures. There is extensive literature available supporting the use of these devices for arterial access site closure, showing reduced time to hemostasis, earlier ambulation and reduced length of hospital stay in comparison to manual compression which is the traditional approach to achieve access site hemostasis. In contrast, there is not significant evidence supporting the use of these devices for closure of femoral venous access site, partly due to limited use of VCD in cardiac electrophysiology procedures, such as catheter ablation for atrial fibrillation and atrial flutter. Another alternative to manual compression, the Figure of 8 stitch has also been used to achieve vascular closure follow catheter ablation of atrial fibrillation and atrial flutter, however it has not been studied formally.

The aim of this registry is to better understand the 'real-world' utilization of VCD or Figure of 8 stitch(F08S) in cardiac ablation procedures and to understand any potential difference between VCD or F08S and manual compression. The outcomes of interest are vascular access site complication rate, time to ambulation and patient perception of pain and overall satisfaction, which is assessed via a survey. The hypothesis of this registry is that there will be an increased patient satisfaction and decreased rate of vascular and bleeding complications with use of either Perclose Proglide system or Figure of 8 stitch for venous closure post atrial fibrillation ablation and atrial flutter ablation procedures in comparison to standard manual compression.

The design will be a prospective observational registry collecting data on patients who underwent catheter ablation for atrial fibrillation and atrial flutter, including administration of a patient survey.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a catheter ablation procedure (radiofrequency ablation or cryoablation) to treat symptomatic paroxysmal atrial fibrillation or atrial flutter
* Patients willing to participate in a short written survey

Exclusion Criteria:

* Patients undergoing ablation for an arrhythmia other than atrial fibrillation/atrial flutter or who are not candidates for an ablation procedure for treatment of atrial fibrillation/atrial flutter
* Patients who are not able to read or understand the English language
* Patients who had recent access site complications within the same hospitalization
* Patients who have baseline thrombocytopenia (platelet count less than 80) or known coagulopathy (INR > 1.5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a catheter ablation procedure (radiofrequency ablation or cryoablation) to treat symptomatic paroxysmal atrial fibrillation or atrial flutter at Saint Luke's Hospital of Kansas City
Sampling Method: Non-Probability Sample
Enrollment: 434 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjaya Gupta, MD, Principal Investigator — Saint Luke's Health System
Locations (1):
- Saint Luke's Hospital of Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dauerman HL, Applegate RJ, Cohen DJ. Vascular closure devices: the second decade. J Am Coll Cardiol. 2007 Oct 23;50(17):1617-26. doi: 10.1016/j.jacc.2007.07.028. PMID 17950141
- [Background] Koreny M, Riedmuller E, Nikfardjam M, Siostrzonek P, Mullner M. Arterial puncture closing devices compared with standard manual compression after cardiac catheterization: systematic review and meta-analysis. JAMA. 2004 Jan 21;291(3):350-7. doi: 10.1001/jama.291.3.350. PMID 14734598
- [Background] Biancari F, D'Andrea V, Di Marco C, Savino G, Tiozzo V, Catania A. Meta-analysis of randomized trials on the efficacy of vascular closure devices after diagnostic angiography and angioplasty. Am Heart J. 2010 Apr;159(4):518-31. doi: 10.1016/j.ahj.2009.12.027. PMID 20362708
- [Background] Nikolsky E, Mehran R, Halkin A, Aymong ED, Mintz GS, Lasic Z, Negoita M, Fahy M, Krieger S, Moussa I, Moses JW, Stone GW, Leon MB, Pocock SJ, Dangas G. Vascular complications associated with arteriotomy closure devices in patients undergoing percutaneous coronary procedures: a meta-analysis. J Am Coll Cardiol. 2004 Sep 15;44(6):1200-9. doi: 10.1016/j.jacc.2004.06.048. PMID 15364320
- [Background] Schulz-Schupke S, Helde S, Gewalt S, Ibrahim T, Linhardt M, Haas K, Hoppe K, Bottiger C, Groha P, Bradaric C, Schmidt R, Bott-Flugel L, Ott I, Goedel J, Byrne RA, Schneider S, Burgdorf C, Morath T, Kufner S, Joner M, Cassese S, Hoppmann P, Hengstenberg C, Pache J, Fusaro M, Massberg S, Mehilli J, Schunkert H, Laugwitz KL, Kastrati A; Instrumental Sealing of Arterial Puncture Site-CLOSURE Device vs Manual Compression (ISAR-CLOSURE) Trial Investigators. Comparison of vascular closure devices vs manual compression after femoral artery puncture: the ISAR-CLOSURE randomized clinical trial. JAMA. 2014 Nov 19;312(19):1981-7. doi: 10.1001/jama.2014.15305. PMID 25399273
- [Background] Vaitkus PT. A meta-analysis of percutaneous vascular closure devices after diagnostic catheterization and percutaneous coronary intervention. J Invasive Cardiol. 2004 May;16(5):243-6. PMID 15152128
- [Background] Maraj I, Budzikowski AS, Ali W, Mitre CA, Kassotis J. Use of vascular closure device is safe and effective in electrophysiological procedures. J Interv Card Electrophysiol. 2015 Aug;43(2):193-5. doi: 10.1007/s10840-015-0005-5. Epub 2015 Apr 29. PMID 25921347
- [Background] Noguchi T, Miyazaki S, Yasuda S, Baba T, Sumida H, Morii I, Daikoku S, Goto Y, Nonogi H. A randomised controlled trial of Prostar Plus for haemostasis in patients after coronary angioplasty. Eur J Vasc Endovasc Surg. 2000 May;19(5):451-5. doi: 10.1053/ejvs.1999.1071. PMID 10828223
- [Background] Duffin DC, Muhlestein JB, Allisson SB, Horne BD, Fowles RE, Sorensen SG, Revenaugh JR, Bair TL, Lappe DL. Femoral arterial puncture management after percutaneous coronary procedures: a comparison of clinical outcomes and patient satisfaction between manual compression and two different vascular closure devices. J Invasive Cardiol. 2001 May;13(5):354-62. PMID 11385148
- [Background] Aytemir K, Canpolat U, Yorgun H, Evranos B, Kaya EB, Sahiner ML, Ozer N. Usefulness of 'figure-of-eight' suture to achieve haemostasis after removal of 15-French calibre femoral venous sheath in patients undergoing cryoablation. Europace. 2016 Oct;18(10):1545-1550. doi: 10.1093/europace/euv375. Epub 2015 Dec 23. PMID 26705565
- [Background] Abo-Salem E, Miller B, Wexler L, Attari M. Vascular Closure Devices for venous accesses in anticoagulated patients after catheter ablation for Atrial Fibrillation. JACC March 17,2015. Volume 65, Issue 10S.
- [Background] Martin JL, Pratsos A, Magargee E, Mayhew K, Pensyl C, Nunn M, Day F, Shapiro T. A randomized trial comparing compression, Perclose Proglide and Angio-Seal VIP for arterial closure following percutaneous coronary intervention: the CAP trial. Catheter Cardiovasc Interv. 2008 Jan 1;71(1):1-5. doi: 10.1002/ccd.21333. PMID 18098171

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Because this is a registry, there are no randomization procedures. The choice of closure method was chosen by each subject's physicians. The subjects were approached for consent after the procedure.
Groups:
- Figure of 8: Figure of 8 stitch is used for venous closure post atrial fibrillation and atrial flutter procedures
- Manual Compression: Manual compression is used to achieve hemostasis after atrial fibrillation and atrial flutter procedures
- Perclose Device: Perclose Proglide system is used for venous closure post atrial fibrillation and atrial flutter procedures
Period: Overall Study
Arm/Group | Figure of 8 | Manual Compression | Perclose Device
Started | 203 | 156 | 75
Completed | 203 | 156 | 75
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Figure of 8 | Manual Compression | Perclose Device | Total
Number analyzed (Participants) | 203 | 156 | 75 | 434
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.34 (11.0) | 64.51 (11.0) | 66.20 (11.0) | 64.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 58 | 33 | 171
  Male | 123 | 98 | 42 | 263
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Hemostasis
Description: Time to achieve hemostasis measured in minutes
Time Frame: 2 days
Population: There were 434 patients included
Measure: Mean (Full Range); unit: minutes
Arm/Group | Figure of 8 | Manual Compression | Perclose Device
Number analyzed (Participants) | 203 | 156 | 75
minutes | 9 [7 to 12.1] | 20 [15 to 20] | 7 [4 to 10.1]

2. Primary Outcome: Ambulation
Description: Time to ambulate following hemostasis measured in hours
Time Frame: 2 days
Measure: Median (Full Range); unit: Hours
Arm/Group | Figure of 8 | Manual Compression | Perclose Device
Number analyzed (Participants) | 203 | 156 | 75
Hours | 2.2 [1.3 to 3.5] | 6.5 [5.1 to 7.8] | 2.2 [1.4 to 3.5]

3. Primary Outcome: Complications
Description: Number of bleeding and vascular complications
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Figure of 8 | Manual Compression | Perclose Device
Number analyzed (Participants) | 203 | 156 | 75
Participants | 3 | 5 | 3

4. Primary Outcome: Hospital Stay
Description: Length of hospital stay in hours
Time Frame: 2 days
Measure: Median (Full Range); unit: hours
Arm/Group | Figure of 8 | Manual Compression | Perclose Device
Number analyzed (Participants) | 203 | 156 | 75
hours | 29 [26 to 30] | 29 [28 to 30] | 27.5 [25 to 29]

5. Post Hoc Outcome: Perception of Pain
Description: Patient's perception of pain is measured using a 5 point Likert scale, range from 1 to 5 with higher scores indicating higher level of pain
Time Frame: 2 days
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Figure of 8 | Manual Compression | Perclose Device
Number analyzed (Participants) | 203 | 156 | 75
units on a scale | 4 [2 to 5] | 4 [2 to 5] | 4 [2 to 5]

6. Post Hoc Outcome: Patient Satisfaction
Description: Patient satisfaction is measured using a 5 point Likert scale with range from 1 to 5 with higher scores indicating greater patient satisfaction
Time Frame: 2 days
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Figure of 8 | Manual Compression | Perclose Device
Number analyzed (Participants) | 203 | 156 | 75
units on a scale | 5 [4 to 5] | 5 [4 to 5] | 5 [4 to 5]

7. Post Hoc Outcome: Need for Manual Compression
Description: Patient's need for manual compression is expressed as number of patients as a whole number
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Figure of 8 | Manual Compression | Perclose Device
Number analyzed (Participants) | 203 | 156 | 75
Participants | 3 | 4 | 1

8. Post Hoc Outcome: Use of Protamine Sulfate
Description: Use of protamine sulfate is expressed as a whole number
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Figure of 8 | Manual Compression | Perclose Device
Number analyzed (Participants) | 203 | 156 | 75
Participants | 182 | 19 | 2

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Figure of 8 | Manual Compression | Perclose Device
All-Cause Mortality (participants affected / at risk) | 0/203 | 0/156 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/203 | 1/156 | 0/75
Other Adverse Events (participants affected / at risk) | 3/203 | 4/156 | 3/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Figure of 8 (N=203) | Manual Compression (N=156) | Perclose Device (N=75)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — large hematoma at the access site requiring 3 units of blood transfusion
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Figure of 8 (N=203) | Manual Compression (N=156) | Perclose Device (N=75)
Hematoma (Vascular disorders) | 3 (3) | 4 (4) | 3 (3) — Minor hematomas that did not require a blood transfusion

LIMITATIONS AND CAVEATS:
Single Center, non-randomized

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT03546439/Prot_SAP_000.pdf